CLINICAL TRIAL: NCT06083935
Title: Effect of Diosmin/Hespiridin Combination on the Clinical Outcomes in Patients With Polycystic Ovary Syndrome
Brief Title: Evaluation of the Effects of Diosmin/Hespiridin Combination on the Clinical Outcomes in Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Tony, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC#166
Record Dates: First submitted 2023-09-21; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Poly Cystic Ovary Syndrome
MeSH Terms: interventions — Diosmin; Contraceptives, Oral, Combined; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin + Combined oral contraceptive (Active Comparator): Metformin (Glucophage ® 500 tablets twice daily)+ Combined oral contraceptive (standard therapy) (Yassmin ® film-coated tablets 3 mg of drospirenone and 0.03 mg of ethinyl estradiol once daily daily)
  Interventions: Drug: Combined oral contraceptive; Drug: Metformin
- Diosmin /Hesperidin + Combined oral contraceptive (Experimental): Diosmin /Hesperidin (Daflon two tablets 500 mg daily)+ Combined oral contraceptive((Yassmin ® film-coated tablets 3 mg of drospirenone and 0.03 mg of ethinyl estradiol once daily daily)
  Interventions: Drug: Daflon; Drug: Combined oral contraceptive
- Diosmin /Hesperidin +Metformin + Combined oral contraceptive combination (Active Comparator): Diosmin /Hesperidin (Daflon two tablets 500 mg daily) +Metformin (Glucophage ® 500 tablets twice daily) + Combined oral contraceptive combination (Yassmin ® film-coated tablets 3 mg of drospirenone and 0.03 mg of ethinyl estradiol once daily daily
  Interventions: Drug: Daflon; Drug: Combined oral contraceptive; Drug: Metformin

INTERVENTIONS:
Drug: Daflon — Daflon; two film coated tablets 500 mg daily
  Arms: Diosmin /Hesperidin + Combined oral contraceptive; Diosmin /Hesperidin +Metformin + Combined oral contraceptive combination
Drug: Combined oral contraceptive — Yassmin ® film-coated tablets 3 mg of drospirenone and 0.03 mg of ethinyl estradiol once daily daily
Drug: Metformin — Glucophage ® 500 tablets twice daily
  Arms: Diosmin /Hesperidin +Metformin + Combined oral contraceptive combination; Metformin + Combined oral contraceptive

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most prevalent disorders worldwide. Insulin resistance, inflammation and disturbance in sex hormone levels are the main contributing factors of this disease.The majority of studies addressing the status of chronic low-grade inflammation in PCOS have focused on the measurement of C-reactive protein (CRP) followed by stimulation of interleukin 6 (IL-6) and tumor necrosis factor (TNF-alpha).

Daflon 500 mg tablets (containing 90% of diosmin and 10% of hesperidin) is used in patients to treat varicose veins, venous ulcers, hemorrhoids and lymphatic insufficiency. It has anti-diabetic, anti-inflammatory, microcirculatory, and antioxidant effects. So the aim of the work is to investigate the effect of Diosmin/Hesperidin in the management of PCOS through evaluation of Oxidative stress and inflammation, improvement of signs and symptoms through patients' follow-up, improvement of PCOS status by sonography and hormonal levels, measuring of anti-diabetic effect by measuring, fasting insulin, HOMA-IR and measuring the improvement of patient's quality of life by using the women health questionnaire (WHQ).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of PCOS aged in the range from18-40 (premenopausal adults) diagnosed with PCOS according to Rotterdam criteria by an expert gynecologist; (1) oligo-ovulation and/or anovulation (2) Clinical and biochemical hyperandrogenism and (3) polycystic ovaries on ultrasonography

Exclusion Criteria:

* 1-Pregnant and nursing women 2-Menopause women 3-Diabetic patients 4-Adrenal hyperplasia 5-Adrenal Tumor 6-Thyroid dysfunction 7-Women on confounding medications which affect ovarian function

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of the inflammation | 4 months
  Improvement of PCOS status by improvement of the inflammatory markers (IL-6)
Improvement of glycemic index | 4 months
  Improvement of glycemic index by measuring fasting Insulin, HOMA-IR

SECONDARY OUTCOMES:
Improvement of PCOS status levels | 4 months
  Improvement of PCOS status by improvement of signs and symptoms, hormone levels
Improvement of patient's quality of life | 4 months
  Improvement of patient's quality of life by using the women health questionnaire (WHQ)

IPD SHARING:
Plan to Share IPD: No